CLINICAL TRIAL: NCT03106090
Title: Comparison of Enhanced Survivorship Care Plans in a Head and Neck Cancer Clinic to Standard of Care
Brief Title: Studying Survivorship Care Plans in Head and Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to meet accrual goals.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00079937
Record Dates: First submitted 2017-03-29; First posted 2017-04-10 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Head and Neck Cancer
Keywords: survivorship care plan; head and neck cancer; survivorship
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Intervention (group receiving eSCPs) will be compared to 2 control groups: group receiving prior standard of care and standard of care SCP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No SCP Control (No Intervention): Patients returning for early follow-up who did not receive SCP.
- SOC SCP Control (No Intervention): Patients returning for early follow-up who received a standard of care SCP.
- eSCP Intervention (Experimental): Patients currently receiving treatment who will be enrolled to receive an "enhanced" SCP (eSCP) with additional information beyond ASCO guidelines tailored to patient concerns and preferences.
  Interventions: Other: educational materials

INTERVENTIONS:
Other: educational materials — The eSCP includes a treatment summary section, a section detailing follow-up and test recommendations, a section on anticipated and potential side effects, as well as additional information specific to their experience/concerns. They will receive a patient education notebook outlining symptoms and their management that is tailored to those that the subject may be likely to experience during their survivorship care trajectory.
  Arms: eSCP Intervention

SUMMARY:
The study will focus on survivorship care for head and neck cancer patients cared for within Duke Cancer Center clinics. Standardized survivorship care plans (sSCP) are being implemented based on the American Society for Clinical Oncology's criteria. These documents provide a summary of treatment received, and list side effects and follow-up information after cancer treatment. Taking advantage of this transition, the investigator will study three groups of patients: (a) early survivors treated before the sSCP was implemented, (b) early survivors treated after the sSCP was implemented, and (c) current patients who will receive an individualized enhanced SCP (eSCP), which will include additional information tailored to patient preferences. The investigators hypothesize that patients receiving enhanced survivorship care plans will increase their knowledge regarding their health care plan and wellness trajectory; increase their ability to identify the symptoms they most likely can expect as a result of their cancer treatment; and be more likely to engage in conversations with their PCP about healthy behaviors and screening guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Completed treatment for a head or neck cancer at Duke Cancer Center within 4 months of consent OR
* Will complete treatment for a head and neck cancer at Duke Cancer Center within 3 weeks of consent AND
* Able to read and understand English
* Capable of giving informed consent
* Are at least age 18.

Exclusion Criteria:

* incompetent for interview (documented diagnosis of active psychosis or dementia) or unable to provide informed consent as assessed by the interviewer; or too sick to participate, as judged by a member of the research team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Head and Neck Cancer Survivor Knowledge | 5 minutes to complete 3 months after treatment end
  Assesses survivor knowledge of potential cancer or treatment-related symptoms and knowledge of healthy behaviors through the use of the Head and Neck Cancer Survivor Knowledge Scale
Change in Head and Neck Cancer Survivor Knowledge | 5 minutes to complete; measured pre-intervention and 3 months after intervention
  Assesses survivor knowledge of potential cancer or treatment-related symptoms and knowledge of healthy behaviors through the use of the Head and Neck Cancer Survivor Knowledge Scale in intervention group

SECONDARY OUTCOMES:
Distress in head and neck cancer survivors | 5 minutes to complete 3 months after treatment end
  Assesses risk of distress defined within post-traumatic stress after treatment through the use of the PTSD Checklist
Distress in head and neck cancer survivors | 5 minutes to complete 3 months after treatment end
  Assesses distress through the use of the NCCN Distress Thermometer
Change in distress for head and neck cancer survivors | 5 minutes to complete; measured pre-intervention and 3 months after intervention
  Assesses risk of distress defined within post-traumatic stress after treatment through the use of the PTSD Checklist in the intervention group
Change in distress for head and neck cancer survivors | 5 minutes to complete; measured pre-intervention and 3 months after intervention
  Assesses distress through the use of the NCCN Distress Thermometer in the intervention group
Uncertainty in head and neck cancer survivors | 5 minutes to complete 3 months after treatment end
  Assesses uncertainty related to presence of symptoms after cancer treatment through the use of the Mishel Uncertainty in Illness Scale -Survivor/Caregiver form
Change in uncertainty in head and neck cancer survivors | 5 minutes to complete; measured pre-intervention and 3 months after intervention
  Assesses uncertainty related to presence of symptoms after cancer treatment through the use of the Mishel Uncertainty in Illness Scale -Survivor/Caregiver form in the intervention group
Quality of life in head and neck cancer survivors | 5 minutes to complete 3 months after treatment end
  Assesses quality of life in head and neck cancer patients EORTC Quality of Life Questionnaire Head & Neck (QLQ H&N35)
Change in quality of life in head and neck cancer survivors | 5 minutes to complete; measured pre-intervention and 3 months after intervention
  Assesses quality of life in head and neck cancer patients EORTC Quality of Life Questionnaire Head & Neck (QLQ H&N35) in the intervention group
Self-efficacy in head and neck cancer survivors | 5 minutes to complete 3 months after treatment end
  Assesses self-efficacy in cancer patients through the use of the Self-Efficacy Scale
Change in self-efficacy in head and neck cancer survivors | 5 minutes to complete; measured pre-intervention and 3 months after intervention
  Assesses self-efficacy in cancer patients through the use of the Self-Efficacy Scale
Information processing in head and neck cancer survivors | 5 minutes to complete 3 months after treatment end
  Assesses information processing in cancer patients through the use of the EORTC QLQ Information Module (QLQ INFO25)
Change in information processing in head and neck cancer survivors | 5 minutes to complete; measured pre-intervention and 3 months after intervention
  Assesses information processing through the use of the EORTC QLQ Information Module (QLQ INFO25)
Survivorship care plan perceptions in head and neck cancer survivors | 5 minutes to complete 3 months after treatment end
  Using open ended questions during a qualitative interview, survivors will provide their perception of how survivorship care plans were useful or not in their care
Survivorship needs after treatment completion -- primary care provider documentation | 10 minutes to complete documentation review of 6 months of PCP records
  Using a documentation checklist developed by the study team, discussions on survivorship needs when returning to clinic will be assessed with a focus on symptom management or incorporation of healthy behaviors to reduce cancer recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Deborah H Allen, PhD, RN, Principal Investigator — Duke Health
Locations (1):
- Duke Health, Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No